CLINICAL TRIAL: NCT05163626
Title: Combined Aerobic Exercise and Cognitive Training for Alzheimer's Disease Prevention in At-Risk Seniors Estimated by An Exosomal Synaptic Protein Model: Cognition and Exosomal Synaptic Proteins Effects
Brief Title: Combined Aerobic Exercise and Cognitive Training in Seniors at Increased Risk for Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICND20210920
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; aerobic exercise; exosome; synaptic protein; biomarker; prevention; cognitive training
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined aerobic exercise and cognitive training program (Experimental)
  Interventions: Behavioral: Combined aerobic exercise and cognitive training program
- Standard health counseling at baseline (No Intervention)

INTERVENTIONS:
Behavioral: Combined aerobic exercise and cognitive training program — Participants will take part in a combined aerobic exercise and cognitive training program. The program will include moderate cycling exercise and cognitive game resolving at the same time. The tasks will be instructed and supervised by a fitness expert and a trained clinical neuropsychologist.
  Arms: Combined aerobic exercise and cognitive training program

SUMMARY:
The study aims to investigate the effect of a long-term combined aerobic exercise and cognitive training program on cognitive function and blood exosomal synaptic protein levels in seniors at increased risk for Alzheimer's Disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia in people older than 65 years worldwide. The neuropathological changes of AD occur decades before the onset of cognitive impairment, suggesting that early identification and timely intervention may postpone the clinical progress. In addition to its characteristic amyloid β and tau pathology, AD is also marked by synaptic dysfunction. Abnormal synaptic protein levels, such as growth associated protein 43 (GAP43), neurogranin, synaptotagmins, and synaptosome associated protein 25 (SNAP25) have been observed in the brain tissue and cerebrospinal fluid (CSF). Blood neuro-exosomal synaptic proteins have emerged as promising predictors for AD and cognitive decline. Particularly, the investigators previously reported a combination of blood neuro-exosomal protein (GAP43, neurogranin, SNAP25, and synaptotagmin 1) can predict AD 5 to 7 years before the clinical onset.

Both physical exercise and cognitive training have been demonstrated to improve cognitive function in AD and to exert a protective effect against developing dementia in the normal aging population. Furthermore, cognitive stimulation is an established modulator of synaptic plasticity and physical exercise might regulate synapse functional and structural change. However, whether cognitive training and physical exercise can alter exosomal synaptic protein levels and the relationship of biomarker changes to cognitive function in those seniors at increased risk for AD remain unclear.

In this study, the investigators aim to

1. assess the effects of a long-term combined aerobic exercise and cognitive training program on cognitive function and the predictive biomarkers (blood neuro-exosomal synaptic proteins: GAP43, neurogranin, SNAP25, and synaptotagmin 1) in seniors at increased risk of AD with abnormally decreased levels of the biomarkers.
2. determine the relationship of biomarker changes with cognitive function in these people.
3. confirm the predictive value of the blood neuro-exosomal synaptic proteins for AD in a longitudinal setting.

ELIGIBILITY:
Inclusion Criteria:

* Mandarin-speaking subjects.
* Not clinically demented.
* Meeting the cutoff values of MMSE and CDR.
* With low levels of blood neuro-exosomal synaptic proteins (GAP43<1983pg/ml, synaptotagmin 1<431pg/ml, neurogranin<1433pg/ml, SNAP25<448pg/ml)

Exclusion criteria:

* Had major neurologic diagnosis (e.g., Alzheimer's disease, Parkinson's disease, stroke, encephalitis, and epilepsy) or other condition that might impair cognition or confound assessments.
* Had a history of psychotic episodes or had major depression (Hamilton Depression Rating Scale score > 24 points).
* Had severe systemic diseases, such as tumors, cardiovascular or orthopedic disorders that can affect the ability to perform the proposed intervention tasks.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function over time as assessed by the Montreal Cognitive Assessment (MoCA) | baseline time, year 1, year 3, year 5, year 7
  MoCA will be performed to evaluate the cognition of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 30, with higher values indicating better cognition.
Change in cognitive function over time as assessed by Mini Mental State Examination (MMSE) | baseline time, year 1, year 3, year 5, year 7
  MMSE will be performed to evaluate the cognition of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 30, with higher values indicating better cognition.
Change in cognitive function over time as assessed by Clinical Dementia Rating (CDR) | baseline time, year 1, year 3, year 5, year 7
  CDR will be performed to evaluate the cognition of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 18, with higher values indicating worse cognition.
Change in cognitive function over time as assessed by Verbal Fluency Test | baseline time, year 1, year 3, year 5, year 7
  Verbal Fluency Test will be performed to evaluate the semantic memory function of participants at the enrollment and year 1, year 3, year 5, year 7. Participants are asked to produce as many animals as possible within 1 minute. The score is the number of animals, with higher scores indicating better cognition.
Change in cognitive function over time as assessed by Digit Span Test-Forward and Backward | baseline time, year 1, year 3, year 5, year 7
  Digit Span Tests will be performed to evaluate the working memory of participants at the enrollment and year 1, year 3, year 5, year 7. The total scores are twelve for each test, with higher values indicating better cognition.
Change in cognitive function over time as assessed by Trail-Making Test Parts A and B (TMT-A and TMT-B) | baseline time, year 1, year 3, year 5, year 7
  TMT-A and TMT-B will be performed to evaluate the executive function of participants at the enrollment and year 1, year 3, year 5, year 7. Scoring is based on time taken to complete the test (e.g., 35 seconds yielding a score of 35), with lower scores indicating better cognition.
Change in cognitive function over time as assessed by Boston Naming Test (BNT) | baseline time, year 1, year 3, year 5, year 7
  BNT will be performed to evaluate the language function of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 30, with higher values indicating better cognition.
Change in cognitive function over time as assessed by the Rey-Osterrieth Complex Figure Test (ROCF) | baseline time, year 1, year 3, year 5, year 7
  ROCF will be performed to evaluate the visuospatial function and other cognition domains of participants at the enrollment and year 1, year 3, year 5, year 7. Participants are asked to produce a complicated line drawing, with higher scores indicating better cognition.
Change in cognitive function over time as assessed by California Verbal Learning Test (CVLT) | baseline time, year 1, year 3, year 5, year 7
  CVLT will be performed to evaluate the memory function of participants at the enrollment and year 1, year 3, year 5, year 7. Participants are asked to finish immediate recall, delayed recall, and delayed recognition tasks in the test, with higher scores indicating better cognition.

SECONDARY OUTCOMES:
Changes in concentrations of blood neuro-exosomal GAP43 over time | baseline time, year 1, year 3, year 5, year 7
  Concentrations of blood neuro-exosomal GAP43 will be evaluated at the enrollment and year 1, year 3, year 5, year 7, and measured in pg/ml.
Changes in concentrations of blood neuro-exosomal neurogranin over time | baseline time, year 1, year 3, year 5, year 7
  Concentrations of blood neuro-exosomal neurogranin will be evaluated at the enrollment and year 1, year 3, year 5, year 7, and measured in pg/ml.
Changes in concentrations of blood neuro-exosomal SNAP25 over time | baseline time, year 1, year 3, year 5, year 7
  Concentrations of blood neuro-exosomal SNAP25 1 will be evaluated at the enrollment and year 1, year 3, year 5, year 7, and measured in pg/ml.
Changes in concentrations of blood neuro-exosomal synaptotagmin1 over time | baseline time, year 1, year 3, year 5, year 7
  Concentrations of blood neuro-exosomal synaptotagmin1 will be evaluated at the enrollment and year 1, year 3, year 5, year 7, and measured in pg/ml.
The area under curve of the blood neuro-exosomal synaptic proteins (GAP43, neurogranin, SNAP25, and synaptotagmin1) for the accurate diagnosis of AD | up to 7 years
  The area under curve is used to show the ability of the blood neuro-exosomal synaptic proteins (GAP43, neurogranin, SNAP25, and synaptotagmin1) to diagnose AD. The value of area under curve is higher, then the ability of the blood neuro-exosomal synaptic proteins to diagnose AD is stronger.

CONTACTS AND LOCATIONS:
Overall Officials: Longfei Jia, MD,PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia L, Zhu M, Kong C, Pang Y, Zhang H, Qiu Q, Wei C, Tang Y, Wang Q, Li Y, Li T, Li F, Wang Q, Li Y, Wei Y, Jia J. Blood neuro-exosomal synaptic proteins predict Alzheimer's disease at the asymptomatic stage. Alzheimers Dement. 2021 Jan;17(1):49-60. doi: 10.1002/alz.12166. Epub 2020 Aug 10. PMID 32776690
- [Background] Jia L, Quan M, Fu Y, Zhao T, Li Y, Wei C, Tang Y, Qin Q, Wang F, Qiao Y, Shi S, Wang YJ, Du Y, Zhang J, Zhang J, Luo B, Qu Q, Zhou C, Gauthier S, Jia J; Group for the Project of Dementia Situation in China. Dementia in China: epidemiology, clinical management, and research advances. Lancet Neurol. 2020 Jan;19(1):81-92. doi: 10.1016/S1474-4422(19)30290-X. Epub 2019 Sep 4. PMID 31494009
- [Background] Chatzi C, Zhang Y, Hendricks WD, Chen Y, Schnell E, Goodman RH, Westbrook GL. Exercise-induced enhancement of synaptic function triggered by the inverse BAR protein, Mtss1L. Elife. 2019 Jun 24;8:e45920. doi: 10.7554/eLife.45920. PMID 31232686
- [Background] Lopez-Ortiz S, Valenzuela PL, Seisdedos MM, Morales JS, Vega T, Castillo-Garcia A, Nistico R, Mercuri NB, Lista S, Lucia A, Santos-Lozano A. Exercise interventions in Alzheimer's disease: A systematic review and meta-analysis of randomized controlled trials. Ageing Res Rev. 2021 Dec;72:101479. doi: 10.1016/j.arr.2021.101479. Epub 2021 Sep 30. PMID 34601135
- [Background] He Z, Gao Y, Alhadeff AL, Castorena CM, Huang Y, Lieu L, Afrin S, Sun J, Betley JN, Guo H, Williams KW. Cellular and synaptic reorganization of arcuate NPY/AgRP and POMC neurons after exercise. Mol Metab. 2018 Dec;18:107-119. doi: 10.1016/j.molmet.2018.08.011. Epub 2018 Sep 12. PMID 30292523
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936